CLINICAL TRIAL: NCT07022418
Title: Prospective Randomized Pilot Trial of Formoterol in Patients With Diabetic Kidney Disease
Brief Title: Formoterol in Diabetes
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Dialysis Clinic, Inc. (Industry)
Responsible Party: Principal Investigator, Joshua Lipschutz, Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00144030
Record Dates: First submitted 2025-05-21; First posted 2025-06-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Nephropathies; Diabetic Kidney Disease
Keywords: Diabetes
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care Only (No Intervention): Standard of Care Treatment Only
- Formoterol Fumarate + Standard of Care Treatment (Experimental): Formoterol Fumarate Inhalation Solution as one 20 mcg unit-dose vial administered twice daily (morning and evening) by nebulization (in addition to standard of care treatment)
  Interventions: Drug: Formoterol furmarate (20 μg)

INTERVENTIONS:
Drug: Formoterol furmarate (20 μg) — Investigators chose to use the long-acting β2-AR agonist, formoterol, because of its efficacy and safety profile in patients with COPD and because formoterol showed the most association with protection from progression of CKD in our retrospective study.
  Arms: Formoterol Fumarate + Standard of Care Treatment

SUMMARY:
The purpose of the study is to evaluate if formoterol fumarate is effective in treating patients with diabetic kidney disease. Study participants will be randomly assigned to either receive formoterol fumarate (in addition to their current standard of care treatment) or standard of care treatment only. Study participants will have a 50% chance of receiving formoterol fumarate and a 50% chance of not receiving formoterol fumarate. Both groups will continue their standard of care treatment during the study. The primary goal is to gather data on feasibility and effect sizes to properly power a future clinical trial.

DETAILED DESCRIPTION:
Glomerular function is highly dependent on specialized cells known as podocytes, which are critical components of glomeruli. Diseases affecting podocytes and the glomerulus, such as diabetes, are the leading causes of ESKD, and there are no specific therapies that restore injury-induced loss of podocyte structure and function. It was previously shown using mouse models of podocyte injury that formoterol fumarate, a long-acting β2-AR agonist given four hours following injury, when glomerular dysfunction is already established, restored glomerular structure, significantly reduced proteinuria, and accelerated recovery of glomerular function. To determine if a similar effect occurred in CKD, specifically DN, investigators used streptozotocin, a murine model of type 1 diabetes, and a high fat diet (HFD), a murine model of type 2 diabetes, to examine the role of formoterol fumarate in DN. Following formoterol fumarate treatment, there was a marked recovery from and reversal of DN in the streptozotocin and HFD mice treated with formoterol fumarate compared to those treated with vehicle alone at the ultrastructural, histological, and functional levels. Investigators also performed a competing risk regression in Veterans aged 65 or over with incident CKD stage 4 to compare the rate of ESKD progression in Veterans without and with COPD, who use β2-AR agonists. Investigators found a 25.6% reduction in the rate of ESKD in Veterans with COPD compared to those without4. In a second cohort of Veterans, Investigators demonstrated significantly slower progression from CKD stage 3 to CKD stage 5 in patients with COPD compared to those without COPD. Together these data indicate that β2-AR agonists, especially formoterol fumarate, may be a novel treatment for DN.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75
* Diagnosis of type 2 diabetes according to American Diabetes Association (ADA) criteria
* On stable medical therapy for at least 3 months
* Stage CKD G2 to G3b; A2-A3 as defined by eGFR with no requirement for renal biopsy for diagnosis
* Diabetic kidney disease as per Nephrologist
* Urinary albumin to creatinine excretion rate (UACR) 200-5000 mg/g/24hrs on at least two occasions (one of these can be a spot UACR)
* HbA1c <8%
* Receiving stable doses of ACE inhibitor or ARB therapy prior to screening (at least 3 months, unless contraindicated) and/or a stable dose of an SGLT inhibitor (at least 3 months preceding enrollment)
* Receiving stable doses of all additional anti-HTN medications, insulin, oral and injectable non-insulin agents and cholesterol lowering medications at least 3 months prior (unless contraindicated) to randomization and agree to maintain until the study's conclusion.
* Willing and able to comply with schedule of events and protocol requirements, including written informed consent.

Exclusion Criteria:

* Female subjects who are pregnant or breast feeding or who plan on becoming pregnant
* Currently take beta-agonists
* Organ transplant recipients
* Any history of New York Heart Association (NYHA) class III/IV heart failure or recent history of serious heart problem (CABG, stroke, MI) in the past 12 months
* Any history of asthma
* Patients with serum potassium levels <3.5 mEQ/L
* Patients with uncontrolled HTN SBP >150mmHg, DBP >95mmHg
* EKG showing QTc elongation or tachyarrhythmia; including sinus tachycardia >100bpm
* Contraindications to formoterol fumarate (hypersensitivity, including patients with known hypersensitivity to ACE inhibitors or ARBs)
* Advanced organ failure
* Untreated/uncontrolled cardiovascular, pulmonary, or gastrointestinal disease
* Patients with BMI >50
* Active untreated cancer
* Alcohol or drug abuse in the past 6 months
* Being involuntarily incarcerated
* Participating in another interventional study
* Unable or unwilling to do the 36-week intervention

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility: refusal rate and adherence during the 36-week treatment | 36 weeks
  The primary measures of feasibility will be study refusal rate and adherence during the 36-week treatment. Refusal rate will be the percentage of individuals who are offered the opportunity to enroll but choose not to accept it. Adherence will be defined as the proportion of doses taken during the 36-week treatment period. For patients who fail to complete the study, adherence will be estimated as the number of doses they report taking for visits at which they are present over the total number of doses they should have received.
To assess the safety, tolerability, and acceptability of the intervention with formoterol | 36 Weeks
  Rates of adverse events and safety measures will be compared between groups. The investigators will assess adherence with the intervention and study medication.
To perform preliminary efficacy testing and determine the variability of albuminuria | 36 Weeks
  Changes in albuminuria will be compared between groups to provide preliminary efficacy testing.
To perform preliminary efficacy testing and determine the variability of eGFR. | 36 Weeks
  Changes in eGFR will be compared between groups to provide preliminary efficacy testing. eGFR will be assessed using the CKD-Epi Formula.

SECONDARY OUTCOMES:
Safety Monitoring: Body Weight | 36 Weeks
  Body weight will be measured using a digital scale accurate to +/- 0.1 kg at Screening, Week 0, Week 24, and Week 36. The investigator monitors changes in participants' body to detect any changes that may indicate treatment effects or safety concerns.
EKG Evaluations | 40 Weeks
  An EKG will be performed at Screening, Week 0, Week 4, Week 16, Week 36, and Week 40. The investigators will be monitoring for new EKG changes suggestive of beta-adrenergic use such as flattening of the T wave, prolongation of the QTc interval, and ST segment depression, and/or serum potassium <3.0 mEQ/L refractory to medical therapy.
Adherence | 36 Weeks
  Adherence will be defined as the proportion of doses taken during the 36-week treatment period. For patients who fail to complete the study, adherence will be estimated as the number of doses they report taking for visits at which they are present over the total number of doses they should have received
Adverse Events | 40 Weeks
  Rate of protocol related adverse events and serious adverse events will be compared between groups
Tolerability and acceptability | 32 Weeks
  Intervention Tolerability: Participants will be asked every four weeks (Week 4-36) to rate on a 1-10 Likert scale how tolerable the intervention was over the past four weeks.
  Intervention Acceptability: Satisfaction with the intervention will be assessed every 4 weeks (Week 4-36) with a questionnaire that asks participants to rate on a 1-10 Likert scale how satisfied they were with specific domains of the intervention over the past 4 weeks. The major domains that will be assessed are satisfaction with: 1) how hard was it to adhere to prescribed treatment, and 2) how likely they feel they can adhere to the prescribed treatment for the next four weeks. Participants will also be asked in open-ended fashion to provide feedback on each domain of the intervention. The investigators will also assess intervention acceptability by comparing the frequency of protocol related adverse events, requirement for protocol modification, and attrition between groups.
Liver Ultrasound Elastography | 36 Weeks
  non-invasive liver ultrasound elastography to determine if the patients had an improvement in liver steatosis with formoterol
Laboratory Evaluations: HbA1c | 40 Weeks
  HbA1c assessments at Screening, Week 0, Week 16, Week 36, and Week 40 will be estimated and compared between and within groups.
Laboratory Evaluations: CMP | 40 Weeks
  Comprehensive Metabolic Panel (CMP) (including hypokalemia assessments) at Screening, Week 0, Week 4, Week 12, Week 24, Week 36, and Week 40 will be estimated and compared between and within groups.
Laboratory Evaluations: Urine Albumin | 40 Weeks
  Change in albuminuria between groups from baseline to the end of the study
Laboratory Evaluations: eGFR | 40 Weeks
  Change in estimated glomerular filtration rate (eGFR, CKD-Epi eGFR formula) between groups from baseline to the end of the study
Safety Monitoring: Heart Rate | 40 Weeks
  The investigator monitors changes in participants' heart rate throughout the trial to detect any changes that may indicate treatment effects or safety concerns.
Safety Monitoring: Blood Pressure | 40 Weeks
  The investigator monitors changes in participants' blood pressure throughout the trial to detect any changes that may indicate treatment effects or safety concerns. Blood pressure (BP) will be measured with a sphygmomanometer (average of 2 seated values taken after five minutes of rest).
Safety Monitoring: Respiratory Rate | 40 Weeks
  The investigator monitors changes in participants' respiratory rate throughout the trial to detect any changes that may indicate treatment effects or safety concerns.
Safety Monitoring: Temperature | 40 Weeks
  The investigator monitors changes in participants' temperature throughout the trial to detect any changes that may indicate treatment effects or safety concerns.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Lipschutz, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States